CLINICAL TRIAL: NCT01030614
Title: Dexamethasone Improves Postoperative Symptoms in Patients Undergoing Elective Laparoscopic Cholecystectomy: A Randomised Clinical Trial.
Brief Title: Dexamethasone Improves Postoperative Symptoms After Laparoscopic Cholecystectomy
Acronym: dxt
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Alejandro Gonzalez-Ojeda, M.D., Ph.D., Full-time Surgical Researcher, Specialties Hospital. Mexican Insitute of Social Security
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Dxt-2009-01
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-01

CONDITIONS: Postoperative Nausea and Vomiting; Postoperative Pain; Postoperative Fatigue
Keywords: Laparoscopic cholecystectomy,postoperative symptoms
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone group (Active Comparator): One hundred five patients were randomized to receive intravenous dexamethasone (8 mg) before laparoscopic cholecystectomy
  Interventions: Drug: Dexamethasone
- Placebo group (Placebo Comparator): One hundred five patients were randomized to receive intravenous placebo before laparoscopic cholecystectomy
  Interventions: Drug: Dexamethasone; Drug: placebo

INTERVENTIONS:
Drug: Dexamethasone — intravenous dexamethasone 8 mgr before laparoscopic cholecystectomy or intravenous placebo before laparoscopic cholecystectomy
Drug: placebo — One hundred five patients were randomized to receive intravenous placebo before laparoscopic cholecystectomy
  Arms: Placebo group

SUMMARY:
Dexamethasone has been reported to reduce postoperative nausea and vomiting (PONV) after laparoscopic cholecystectomy (LC). However, its effects on other surgical outcomes such as pain and fatigue have been unclear. We evaluated the efficacy of preoperative dexamethasone in ameliorating postoperative symptoms after LC.

Methods: Prospective, double-blind, placebo-controlled study, 210 patients scheduled for elective LC were analyzed after randomization to intravenous dexamethasone (8 mg) or to a placebo. All patients underwent standardized procedures for general anesthesia and surgery. Episodes of PONV and pain and fatigue scores were recorded on a visual analogue scale. Analgesic and antiemetic requirements were also recorded.

DETAILED DESCRIPTION:
Patients and methods

Patients Between January 2007 and August 2008, 210 patients undergoing LC were studied in accordance with a prospective, randomized, double-blind clinical trial. Patients were randomized to receive intravenous dexamethasone (8 mg) or homologated placebo 60 minutes before skin incisions, using an equal number of blind envelopes. Patients of American Society of Anesthesiologists (ASA) classes III and IV were excluded. Further exclusion criteria were age more than 80 years; pregnancy; treatment with steroids; severe diabetes mellitus (HbA1c > 8%); use of opioids, sedatives or any kind of analgesics less than one week before LC; a history of alcohol or drug abuse; preoperative diagnosis of acute cholecystitis, acute pancreatitis, choledocolithiasis, gallbladder carcinoma and/or conversion of the LC to an open procedure. All patients were followed from hospital admission until 30 days after the surgical procedure.

Anesthesia and surgery All patients underwent a standardized general anesthesia procedure. Induction used intravenous midazolam (1.5 mg) and fentanyl (3-5 mcg/kg of body weight) and propofol (2 mg/kg body weight). Anesthesia was maintained with 2 to 3% sevoflurane and 100% oxygen concentration. Neuromuscular blocking was maintained with intravenous vecuronium (0.1 mg/kg body weight). All patients were monitored with indirect determinations of arterial pressure and heart rate using the standard technique as well as expired CO2 content and oxygen blood saturation. A nasogastric tube was placed in all patients during the operation and taken out at the end of the surgical procedure. Afterwards, all patients were extubated and transferred to the immediate postsurgical care unit with cardiovascular and oxygen monitoring.

All patients received preoperative intravenous antibiotics (1 g of intravenous first-generation cephalosporin). LC was performed using a 2-handed, 4-trocar technique with 2 10-mm ports and 2 5-mm ports. A 10-mm subumbilical port was introduced by the open method, subsequently creating a pneumoperitoneum, maintained at 12 to 14 mmHg of intra-abdominal pressure. All of the laparoscopic treatments were performed by expert surgeons, each having sufficient experience of laparoscopic surgery (more than 150 LCs per year). The skin was closed with single nonabsorbable sutures. Closed suction drains were placed in the inferior surface of the liver, using a 5-mm lateral port in some patients according to each surgeon's preference. The drains were removed during the following 12-24 h.

Analgesia and antiemetics Pain and fatigue were assessed preoperatively and immediately on return to the recovery room, and at 6, 12 and 24 h after the operation using a visual analogue scale (VAS; 0 = no pain/fatigue to 10 = most severe pain/fatigue) [7,15,16]. Analgesia was given as intravenous sodium ketorolac (30 mg every 8 h). Intramuscular buprenorphine (0.15-0.30 mcg) was used as a backup analgesic medication. The incidence of PONV was recorded immediately on return to the recovery room and at 6, 12 and 24 h, after the operation, using a four-point ordinal scale (0 = none, 1 = nausea, 2 = nausea with request for antiemetic, 3 = vomiting). Intravenous ondansetron (4-8 mg) was given for antiemetic treatment on demand.

Data collection and statistical analysis Postoperative complications were recorded during hospitalization and the patients were followed up to 30 days after discharge. Data collected also included patient age, sex, body mass index (BMI), ASA score, history of previous abdominal surgery, anesthesia and operation time and frequency of use of analgesic and antiemetic drugs. These parameters were summed and compared between the dexamethasone and placebo groups. The study endpoints were degree of postoperative nausea, vomiting, pain and fatigue and additional analgesic and antiemetic drugs.

The sample size was predetermined. We expected a 20% difference in the incidence of nausea and vomiting between groups. The error alpha error was set at 0.05 and beta error at 0.20; n = 103 patients for each group was considered adequate, according to a power analysis. Results were expressed as percentages and as the mean ± standard deviation (SD). Student's t test and the chi squared test were used for the analysis of quantitative and qualitative data, respectively. Differences were considered statistically significant at p < 0.05.

Ethical considerations The study was conducted according to the principles of the Declaration of Helsinki of 1989 and the Mexican Health Guidelines. The Ethical and Research Committees of the Regional Hospital # 110 of the Mexican Institute for Social Security in Jalisco, Mexico approved all protocols. Full, written informed consent was obtained from all patients before their inclusion in the study.

ELIGIBILITY:
Inclusion Criteria: Adult patients (ASA I and II) with symptomatic cholelithiasis.

Exclusion Criteria:Patients of American Society of Anesthesiologists (ASA) classes III and IV were excluded. Further exclusion criteria were age more than 80 years; pregnancy; treatment with steroids; severe diabetes mellitus (HbA1c > 8%); use of opioids, sedatives or any kind of analgesics less than one week before LC; a history of alcohol or drug abuse; preoperative diagnosis of acute cholecystitis, acute pancreatitis, choledocolithiasis, gallbladder carcinoma and/or conversion of the LC to an open procedure.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2007-01; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
postoperative nausea and vomiting after elective laparoscopic cholecystectomy | At recovery room after laparoscopic cholecystectomy and after 6, 12 and 24 hours. Follow-up during 30 days after surgery

SECONDARY OUTCOMES:
Pain and postoperative fatigue | At recovery room after laparoscopic cholecystectomy and after 6, 12 and 24 hours. Follow-up 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Gonzalez-Ojeda, M.D., Ph.D., Principal Investigator — Full-time Surgical Researcher and Professor of Surgery. Surgical Research Unit. Specialties Hospital. Mexican Institute of Social Security. Guadalajara, Jal. Mexico
Locations (1):
- Department of Surgery and Department od Anesthesiology. Specialties Hospital. Westerm Medical Center, Mexican Institute of Social Security., Guadalajara, Jalisco, Mexico